CLINICAL TRIAL: NCT03907761
Title: Hydrodissection of Recurrent Laryngeal Nerve: Case Series
Status: Completed | Type: Observational
Sponsor: Ankara University (Other)
Responsible Party: Principal Investigator, Serkan Akbulut, Principal Investigator, Ankara University
Other Study IDs: 06-480-19
Record Dates: First submitted 2019-04-03; First posted 2019-04-09 (Actual); Last update posted 2019-04-09 (Actual); Status verified 2019-04

CONDITIONS: Recurrent Laryngeal Nerve Injuries
Keywords: thyroidectomy; recurrent laryngeal nerve; hydrodissection
MeSH Terms: conditions — Recurrent Laryngeal Nerve Injuries

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Hydrodissection — high velocity stream of normal saline is given to the dissection area by help of 10 ml syringe

SUMMARY:
This study evaluates the hydrodissection technique in recurrent laryngeal nerve (RLN) dissection in thyroid surgeries. In this study hydrodissection of RLN was performed routinely in thyroid surgeries.

DETAILED DESCRIPTION:
Thyroid surgery is one of the most frequently performed surgical procedures. Recurrent laryngeal nerve (RLN) injury is the most annoying complication of thyroid surgery. According to literature 0.5-5% and 1-30% of patients is reported to have permanent or temporary RLN injury after the surgery, respectively.

RLN innervates all intrinsic muscles of larynx with the exception of cricothyroid muscle. Injury of RLN causes vocal cord paralysis. Unilateral RLN injury causes hoarseness, but when RLNs are bilaterally damaged aspiration during swallowing or life threatening dyspnea can occur according to severity of glottal narrowing.

Hydrodissection is described in laparoscopic cholecystectomy, cataract surgery, carpal tunnel syndrome treatment where meticulous dissection must be carried out as mentioned above. This technique helps exploring anatomical landmarks by gentle dissection without giving harm to tissues. In thyroid surgery hydrodissection is performed to dissect foamy planes and increase visualization of RLN by high velocity stream of warm saline. Despite being used extensively in routine clinical practice to our best knowledge no report evaluating hydrodissection in thyroid surgery exists in the literature up to date.

In this study, investigators aimed to assess the incidence of RLN damage observed in our series by hydrodissection of RLN during thyroid surgery.

To prevent RLN damage, a good knowledge of anatomy and surgeon's experience are crucial. Routine visualization of RLN along tracheoesophageal sulcus, following the course of RLN near suspensory ligament of berry ligament until entering the larynx is recommended to avoid RLN injury. But still some surgeons declare that visualization of RLN is not possible in all operations. Therefore staying close to thyroid capsule during thyroidectomy is considered to be a good surgical practice to preserve the nerve.

Accurate knowledge of RLN anatomical variations, RLN landmarks such as relation of the nerve with inferior thyroid artery branches, berry ligament, inferior horn of thyroid cartilage during thyroidectomy, is essential as mentioned in the literature. Also inflammatory processes of thyroid (thyroiditis), large nodules, previous operations can change the course of nerve. Hence meticulous dissection of RLN should be performed. In simple thyroidectomies lateral or inferior dissection of RLN is the most common approach but in challenging cases such as large nodules, plunging thyroid gland, neck extension limitations, superior approach, craniocaudal dissection of RLN is accepted to be more appropriate . In our study, both lateral and superior approach were used, hydrodissection of foamy tissue and visualization of the nerve by removing blood and debris via high velocity stream of saline was the main point.

Today, various methods of nerve monitoring and stimulation techniques are in use. Intraoperative nerve monitoring (IONM) significantly reduces iatrogenic RLN injury, helps identification of nerve especially in cases with anatomical variations and points early warning of nerve injury. But disadvantages of IONM like improper electrode position leading to nerve damage must be kept in mind. In the study investigators used IONM in only one case which had a story of RLN injury at the previously operated site. Hydrodissection of RLN is also helpful in use of IONM by allowing dissection of the planes gently just like the gas does in laparoscopy. In our country, since government does not pay for it, investigators cannot use IONM routinely. However hydrodissection is an easily applicable, non time-consuming and cheap technique.

In this study consecutive patients underwent thyroidectomy for various thyroid diseases by one surgeon were included in the study. All the patients' demographic variables (age, sex), operation type (bilateral total thyroidectomy, hemithyroidectomy (total lobectomy and isthmectomy), completion total thyroidectomy, whether central neck compartment dissection was performed), pathology reports, nerves at risk were noted retrospectively. RLN exploration was routinely done to avoid nerve damage on the resected lobe side. Hydrodissection technique was performed while exploring RLNs differently from routine thyroidectomies. For hydrodissection a 10 ml syringe was used with a needle of 1 cm length. After ligation of middle thyroid vein and superior thyroid vessels, the thyroid lobe gently retracted medially and carotid arter laterally by retractors, hydrodissection was performed by high velocity stream of warm-normal saline to the foamy dissection area of RLN and berry ligament (Ethical approval was obtained).RLN detection and dissections were performed with hydrodissection. High velocity stream of normal saline is given to the dissection area by an 10 ml syringe. This dissected all the planes in the field like gas insufflation does in laparoscopic surgery . This technique helped RLN dissection without giving harm to any tissue and nerve itself. RLN integrity was checked by mobility of vocal cords 3 days prior to surgery, postoperative 3. day of surgery and if any movement change deteceted at postoperative 3. day, also reevaluation was made 1 month after the surgery. Also during extubation after operation completed, vocal cord movements are checked by direct visualization.

ELIGIBILITY:
Inclusion Criteria:

*patients undergoing thyroidectomy for various thyroid diseases

Exclusion Criteria:

* patients in whom RLN palsy detected by indirect laryngoscopy before surgery

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: all the patients undergoing to thyroidectomy for thyroid nodules
Sampling Method: Non-Probability Sample
Enrollment: 34 (Actual)
Dates: Start 2016-02-01 (Actual); Primary Completion 2017-08-31 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
mobility of vocal cords preoperative to thyroid surgery | 3 days before surgery
  to assess if there is RLN palsy prior thyroidectomy operation preoperative evaluation of vocal cords by indirect laryngoscopy were performed 3 days prior to surgery routinely.

SECONDARY OUTCOMES:
mobility of vocal cords at the postoperative 3. day | 3 days after thyroidectomy
  to evaluate the RLN injury after thyroidectomy with hydrodissection operation, at the postoperative 3. day, vocal cord damage was evaluated with indirect laryngoscopy
mobility of vocal cord at the injured side | 1 month after the operation
  if there was a RLN damage after the operation detected by indirect laryngoscopy at postoperative 3. day, vocal cord movement at the injured side will be reevaluated by indirect laryngoscopy

IPD SHARING:
Plan to Share IPD: No